CLINICAL TRIAL: NCT05122585
Title: Magnetic Tracer in the Sentinel Node Procedure in Breast Cancer: the Non-radioactive Alternative for Radio-isotopes
Acronym: MagTrace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Collaborators: Sysmex America, Inc. (Industry)
Responsible Party: Principal Investigator, Yvonne Vissers, Principal investigator, Zuyderland Medisch Centrum
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METCZ20200211
Record Dates: First submitted 2021-11-04; First posted 2021-11-17 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: MagTracer; Sentinel Lymph Node; Breast Cancer; MagSeed; Magnetic Tracer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective MagTrace patients (Experimental): All prospective patients will receive a MagSeed in the diagnosed breast cancer tumor. In addition, they will receive MagTrace to detect the sentinel lymph node during surgery. Since this is an experimental study, the patients will also be injected with the golden standard of Technetium tracer.
  Interventions: Procedure: MagSeed and MagTrace in breast cancer patiënts

INTERVENTIONS:
Procedure: MagSeed and MagTrace in breast cancer patiënts — Combining MagSeed and Magtracer to perform a wide local excision breast conserving surgery and sentinel node biopsy.

SUMMARY:
Rationale:

In breast cancer, a sentinel node procedure is performed to investigate whether malignant cells have spread to the axillary lymph nodes. This is an important part of determining the stage of breast cancer and the final treatment plan.

A disadvantage of the sentinel node procedure is that it is performed using radioactive tracing with concomitant radiation exposure for the patients and involved health care personnel. In addition, the use of radioactive tracing puts high demands on the logistics in the operation theatre: the capacity of patients that can be treated in one day is limited and the radio-active tracing leads to many time-consuming precautionary measures.

A radiation free alternative would therefore have multiple advantages. Not only with respect to radiation exposure for the patients and health care workers, but also by reducing the waiting time for operation for the patients as it will make the planning of patients for surgery more efficient.

Recently, a radiation free tracer for the sentinel node procedure has become available (Magtrace). This tracer has been tested in small-case studies and is currently used as standard care in several hospitals around the world.

Objective:

The primary objective of this study is to evaluate the diagnostic accuracy of Magtrace in the sentinel node procedure in breast cancer in the Breast Care Centre in Zuyderland Medical Centre; with the ultimate goal to make the sentinel node procedure a radiation free process.

Study design:

A prospective cohort of forty patients with breast cancer and an indication for a sentinel node procedure will be injected with both Technetium (radioisotope) and Magtrace (magnetic). All patients in this study will receive both tracers.

Study population:

Patients of 18 years or older with breast cancer and an indication for a sentinel node procedure will be included. These patients will be recruited by their breast surgeon in the outpatient department of the Breast Care Centre in Zuyderland Medical Centre.

Intervention (if applicable):

Sentinel node procedure using a magnetic tracer next to Technetium.

Main study parameters/endpoints:

The concordance in detection of sentinel nodes by Magtrace and the Technetium tracer, measured by the sensitivity and specificity of Magtrace in detecting sentinel nodes with Technetium tracer as gold standard.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The goal of this project is evaluating the diagnostic accuracy of Magtrace in the sentinel node procedure. To establish that Magtrace is a non-inferior and a non-radioactive alternative for Technetium with respect to reliability in detecting metastases. The ultimate goal is to make the sentinel node procedure a radiation free process.

ELIGIBILITY:
Inclusion Criteria:

* Female patient of 18 years or older.
* Patient with breast cancer and indication for sentinel node procedure.

Exclusion Criteria:

* Patients with a previous history of the sentinel node procedure or axillary lymph node dissection in the unilateral breast.
* Unable to comprehend implications and extent of study and sign for informed consent.
* Known allergy or hypersensitivity to iron oxide or dextran.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
The concordance in detection of sentinel nodes by Magtrace and the Technetium tracer. | During surgery
  Number of sentinel lymph nodes detected using MagTrace and Technetium and their concordance.

SECONDARY OUTCOMES:
Operation time sentinel node procedure | During Surgery
  Surgery time.

CONTACTS AND LOCATIONS:
Locations (1):
- Zuyderland Medical Center, Sittard, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No